CLINICAL TRIAL: NCT07127263
Title: Comparison of Longer Term Outcomes Following the LungCast "Smoking Cessation in Lung Cancer Study". Revisiting the Original LungCast Research Cohort to Look at Longer-term Outcomes (5+ Years) in Newly Diagnosed Lung Cancer, Within Hywel Dda University Health Board Participants Only, Who Were Smokers, Ex-smokers, Never Smoker and Quitters.
Brief Title: Comparison of Longer-term (5 Year+) Outcomes (Survival) of Smokers, Ex-smokers, Never Smoker and Quitters
Acronym: LungCast2
Status: Completed | Type: Observational
Sponsor: Hywel Dda Health Board (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 339817
Record Dates: First submitted 2025-05-07; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer - Non Small Cell Squamous
Keywords: Smoking cessation; Lung cancer; Survival; Tobacco
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnosed Lung Cancer: Patients diagnosed with Lung Cancer, with smoking status recorded at time of diagnosis.

SUMMARY:
Between 2010-2020, the LungCAst observational study followed 3700 patients newly diagnosed with lung cancer across 33 hospitals in Wales and England for 2 years to see if smoking status at time of diagnosis predicted survival rate. This research was sponsored and led by Hywel Dda University Health Board (HDUHB).

This new study examines the health records, (of only the HDUHB participants included in the original LungCAst study), over a longer period of time to see if the benefits of stopping smoking at point of diagnosis with lung cancer continues over a longer period of time (5 years+).

DETAILED DESCRIPTION:
A study into longer-term outcomes from the LUNGCAST study: comparing survival and healthcare utilisation according to smoking status in people with lung cancer, beyond 2 years. By obtaining Hospital Episode Statistics (HES) extract from the Welsh Patient Administration System (WPAS) and Welsh Clinical Portal (WCP) the investigators can retrospectively follow the cohort participants over time and analyse health care utilisation activity, using univariate and multivariate analysis on the effect of smoking status on survival. The Kaplan-Meier method, will be used to estimate the probability of survival over time.

ELIGIBILITY:
Inclusion Criteria:

All patients from the Hywel Dda University Health Board's(HDUHB) site that participated in the original LungCast study

Exclusion Criteria:

* Individuals that did not participate in the original LungCast study in the HDUHB site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Hywel Dda University Health Board's (HDUHB) site that participated in the original LungCast study.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Comparison of longer-term (5 year+) outcomes (survival) of smokers, ex-smokers and never smokers diagnosed with lung cancer between 2010 and 2020 | From date of diagnosis (of having lung cancer) for 5 years
  Following participants with lung cancer over a 5 year period, by reviewing ongoing healthcare activity via HES extraction and applying the Kaplan-Meier method, to evaluate if smoking status at diagnosis predicts better survival rates over a longer period of time. Univariate and multivariate analysis on the effect of smoking status on survival will also be applied.

CONTACTS AND LOCATIONS:
Locations (1):
- Hywel Dda University Health Board, Carmarthen, Carmarthenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided